CLINICAL TRIAL: NCT02237703
Title: Kappa Opioid Receptor Imaging in Post-traumatic Stress Disorder (PTSD)
Status: Terminated | Type: Observational
Why Stopped: The original PI, Alexander Neumeister, left NYULMC. No data was analyzed.
Sponsor: NYU Langone Health (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: S12-01521
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Post-traumatic Stress Disorder (PTSD); Trauma
Keywords: Post-traumatic Stress Disorder (PTSD); Positron emission tomography (PET); Neuroimaging; Kappa opioid receptor (KOR)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Post-traumatic stress disorder (PTSD): Post-traumatic stress disorder (PTSD)
  Interventions: Other: Positron emission tomography (PET) imaging
- Trauma Control (TC): Trauma Control (TC)
  Interventions: Other: Positron emission tomography (PET) imaging
- Healthy Control (HC): Healthy Control (HC)
  Interventions: Other: Positron emission tomography (PET) imaging

INTERVENTIONS:
Other: Positron emission tomography (PET) imaging — Positron emission tomography (PET) imaging

SUMMARY:
This study uses positron emission tomography (PET) imaging to measure kappa opioid receptors (KOR) in the brains of individuals with and without post-traumatic stress disorder (PTSD). The investigators propose to recruit 45 drug-naïve individuals, N=15 patients with PTSD, N=15 trauma-exposed, but asymptomatic healthy control subjects (TC) and N=15 non-trauma exposed healthy control subjects (HC) to participate in one magnetic resonance imaging (MRI) and one PET study. The investigators will also carefully document trauma history, and collect behavioral and neuroendocrine measures to provide a more integrative view on the neurobiology of PTSD and its phenotype. The investigators predict PTSD will show greater carbon - 11 (11C)[11C]LY2795050 volume of distribution (VT) (i.e. KOR binding) values than control populations in an a priori defined PTSD circuit.

ELIGIBILITY:
Inclusion criteria for patients with PTSD:

1. age 18-55 years old
2. currently diagnosed with PTSD and symptomatic with a Clinician-Administered PTSD Scale (CAPS) score > 50.

Exclusion criteria for patients with PTSD:

1. any primary Axis I disorder other than PTSD (e.g. psychosis)
2. medical or neurological illnesses likely to affect physiology or anatomy, i.e. uncontrolled hypertension, cardiovascular disorders
3. a history of drug (including benzodiazepines (BZD)) dependence (Diagnostic and Statistical Manual of Mental Disorders (DSM IV) criteria) within 1 year of the study and lasting longer than 2 years, except for alcohol dependence
4. current pregnancy (as documented by pregnancy testing at screening or on the day of PET imaging study)
5. current breast feeding
6. use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day, or cannot abstain from smoking during the prescribed tests
7. acute suicidal ideation or behavior, as defined by suicidal ideation and behavior during the 3-month period prior to enrollment in the study and while being enrolled in the study
8. general MRI exclusion criteria, i.e. pacemakers, metals in the body
9. Human immunodeficiency virus (HIV) (due to possible neuropsychiatric effects);
10. use of opioid medications within 2 weeks of the PET study
11. having an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participation in the study
12. seriously claustrophobic
13. blood donation within 8 weeks prior to the study.

Inclusion criteria for Healthy Subjects:

1. age 18-55 years old
2. no personal or first-degree family history of any Axis I diagnosis.

Exclusion criteria for Healthy Subjects:

1. any history or current primary Axis I disorder
2. medical or neurological illnesses likely to affect physiology or anatomy, i.e. uncontrolled hypertension, cardiovascular disorders
3. a history of drug (including benzodiazepines [BZD]) dependence (DSM IV criteria) within 1 year of the study and lasting longer than 2 years, except for alcohol dependence
4. current pregnancy (as documented by pregnancy testing at screening or on the day of PET imaging study)
5. current breast feeding
6. use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day, or cannot abstain from smoking during the prescribed tests
7. acute suicidal ideation or behavior, as defined by suicidal ideation and behavior during the 3-month period prior to enrollment in the study and while being enrolled in the study
8. general MRI exclusion criteria, i.e. pacemakers, metals in the body
9. HIV (due to possible neuropsychiatric effects)
10. use of opioid medications within 2 weeks of the PET study
11. having an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risks associated with participation in the study
12. seriously claustrophobic
13. blood donation within 8 weeks prior to the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects are between the age range of 18 to 55, are medically healthy and currently not taking any medications to treat any medical illness, have a history of post-traumatic stress disorder, or are a healthy control who has or has not been exposed to trauma.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Volume of distribution (VT) of cerebral KOR expression in PTSD and healthy control subjects with and without trauma history using the KOR radioligand [11C]LY2795050 and PET | Two months
  To examine group differences in cerebral KOR expression in PTSD and healthy control subjects with and without trauma history using the KOR radioligand [11C]LY2795050 and PET.
  Hypothesis: PTSD will show greater [11C]LY2795050 VT (i.e. KOR binding) values than control populations in an a priori defined PTSD circuit.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Marmar, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States